CLINICAL TRIAL: NCT07357701
Title: Identifying Genome Variants and Evaluating PRDM9 and piRNA Clusters as Candidates for Infertility in a Cohort of Individuals With Non-Obstructive Azoospermia (NOA) or Primary Ovarian Insufficiency (POI)
Brief Title: Identifying Genome Variants in Non-Obstructive Azoospermia (NOA) or Primary Ovarian Insufficiency (POI)
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002332; 002332-CH
Record Dates: First submitted 2026-01-21; First posted 2026-01-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Primary Ovarian Insufficiency; Azoospermia; Oligospermia
Keywords: NOA; POI; Premature Ovarian Insufficiency; oligospermia; azoospermia; diminished ovarian reserve; nonobstructive azoospermia; Primary Ovarian Insufficiency; Infertility
MeSH Terms: conditions — Primary Ovarian Insufficiency; Azoospermia; Oligospermia; Azoospermia, Nonobstructive; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non obstructive azoospermia: Men aged 18 and older who have no semen in the ejaculate with no evidence of pathologic transport of sperm
- Oligospermia: Men aged 18 or older who have a concentration less than 5 million/mL in ejaculate with no other known cause of oligospermia.
- Primary ovarian insufficiency: Women who have been diagnosed with primary ovarian insufficiency

SUMMARY:
Background:

Infertility affects 1 in 6 people. Often, the causes of infertility are unknown. Treatments are successful in only about 50% of cases. Infertility caused by non obstructive azoospermia in males and primary ovarian insufficiency in females can have genetic causes. Researchers want to learn more about these genes.

Objective:

To identify genes that may cause infertility.

Eligibility:

Adult men and women with non-obstructive azoospermia (NOA) or primary ovarian insufficiency (POI) of unknown cause.

Design:

Participants will provide a saliva sample. A kit will be sent to their home. The kit will contain a collection tube and a cotton swab. They will swirl the swab inside their mouth and then seal it in the tube. They will mail the tube back to the researchers.

Male participants who are having a procedure done to collect tissue from their testes may opt to have leftover tissue provided to study researchers. This tissue would otherwise have been discarded. No new procedures will be performed just for this study.

Data may be collected from participants medical records.

DETAILED DESCRIPTION:
Study Description:

PRDM9 and the piRNA pathway have well established roles in meiosis and are known to cause infertility in mouse, yet have not been systematically evaluated for a role in human infertility. We will utilize a combination of genome sequencing, targeted PacBio sequencing, and in vitro assays to evaluate these compelling candidates as causative for human infertility. All participants will be asked to provide saliva or blood samples as a source of genomic DNA for sequencing. A small subset of participants who undergo surgery as part of their diagnosis and treatment plan will be asked to consent to research use of leftover testicular biopsies from these procedures.

Objectives:

Primary Objective:

To determine the sequence of PRDM9 and noncoding piRNA clusters in a cohort of individuals with infertility. These loci are inherently unstable in the genome, and we hypothesize that sequence variants in these loci are causative for infertility.

Secondary Objectives:

Identify genome variants in novel or previously reported infertility candidate genes. Genome variants in hundreds of genes have been reported as candidates for infertility, and collective data from additional cohorts is needed to evaluate the gene-disease relationship of these infertility candidate genes.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Adult male or female, of reproductive age
4. Clinical diagnosis of NOA, oligospermia, or POI.
5. In good general health with no medical history suspected as the cause of infertility.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current use of medications that may cause infertility (chemotherapy, etc.)
2. Pregnant or lactating
3. Medical history indicating known common cause of infertility such as karyotype anomalies, Y-chromosome microdeletions, known monogenic causes, or other medical history affecting gamete production (i.e. injuries, surgical operations, infections, radiation, or chemotherapy).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seeking infertility care diagnosed with primary ovarian insufficiency, non obstructive azoospermia, or oligospermia will be offered the opportunity to enroll in genetic sequencing to further evaluate genetic causes of infertility.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Genetic associations with infertility (primary ovarian insufficiency, oligospermia, non obstructive azoospermia) | 5 years
  Across 5 years we will sequence patients with POI and NOA to determine genetic associations with infertility

CONTACTS AND LOCATIONS:
Overall Officials: Todd S Macfarlan, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Shady Grove Fertility, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002332-CH.html